CLINICAL TRIAL: NCT02854670
Title: A Study of the Effects of Topical Capsaicin in the Treatment of Provoked Vestibulodynia
Acronym: CAPSIVU
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P/2013/199
Record Dates: First submitted 2016-08-01; First posted 2016-08-03 (Estimated); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Vestibulodynia
Keywords: capsaicin; pain improvement; provoked vulvodynia
MeSH Terms: conditions — Vulvodynia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Capsaicin patch (Experimental): Cuttable capsaicin patch. 2 patches of 4 cm² (2 x 2cm), for a total of 2.5 mg of capsaicin.
  Interventions: Drug: Capsaicin patch

INTERVENTIONS:
Drug: Capsaicin patch — After a pre-medication with paracetamol, patches are applied and removed after 20 minutes. Patients remain under observation for 2 hours after removal.

SUMMARY:
This study aims to assess the pain on contact in provoked vestibulodynia, measured with Visual Analogic Scale at week 0/week 2/week 6/week 12 after applying a patch of capsaicin.

ELIGIBILITY:
Inclusion Criteria:

* Provoked vulvodynia, rated B2a according to 2003 International Society for the Study of Vulvovaginal Disease (ISSVD) classification
* Pain ≥ 4 on Visual Analogic Scale (VAS)
* Subject refractory to at least 2 conventional treatments (tricyclic antidepressants, anticonvulsants at analgesic doses , biofeedback physical therapy, psychological assessment in a context of chronic pain) or to botulinum toxin A
* If a former treatment with botulinum toxin A was performed: patient must be in treatment failure (= no decrease over 50% of the pain 3 months after initiation of the treatment)
* Negative screening test results
* Menopause, surgically sterilized women or women using effective contraceptive method
* Good understanding and predictable adherence to the protocol
* Beneficiary/affiliated to French social security/social healthcare
* Signed Informed Consent Form

Exclusion Criteria:

* Predictable poor adherence
* Pregnant or breastfeeding women
* Diabetes mellitus type 1 or type 2
* Major mental disorders
* Underlying etiology such as chronic vulvar disease
* Initial vulvar erythema
* Vulnerable subjects (particularly adults under guardianship)
* Ongoing medical treatment with tricyclic antidepressants or anticonvulsants at analgesic doses

Subject refractory to conventional treatments (tricyclic antidepressants and benzodiazepines doses analgesics, physiotherapy type of biofeedback)

Good understanding and predictable adherence to the protocol beneficiary/affiliated to French social security/social healthcare signed Informed Consent Form

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-01-20 (Actual); Primary Completion 2021-02-03 (Actual); Study Completion 2021-02-03 (Actual)

PRIMARY OUTCOMES:
Pain assessment with Visual Analogic Scale (using a q-tip) | week 12
  Assessment of provoked pain with Visual Analogic Scale (using a q-tip)

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Pelletier, MD, Principal Investigator — CHU Besançon
Locations (1):
- CHU Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No